CLINICAL TRIAL: NCT01630005
Title: Talk Therapy After Stroke. PS-POST AVC
Brief Title: Talk Therapy After Stroke
Acronym: PS-POST AVC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-A00905-34
Record Dates: First submitted 2012-02-20; First posted 2012-06-28 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2010-12

CONDITIONS: Adams-Stokes Syndrome
MeSH Terms: conditions — Adams-Stokes Syndrome | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Talk therapy (Experimental): A cohort of 25 patients
  Interventions: Behavioral: talk therapy

INTERVENTIONS:
Behavioral: talk therapy — Psychotherapy

SUMMARY:
Strokes are the first cause of acquired physical disability among adults. Some studies proved that depression is often an unrecognized complication from stroke, associated with a vital prognosis, functional and cognitive pejorative diagnosis. It led us to pose the hypothesis of the existence of a particular psychological state after stroke particularly favorable to a psychotherapeutic alliance. So, this longitudinal monocentric study aims to estimate the feasibility of a talk therapy and its impact on the anxio-depressive symptomatology after stroke.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or aemoragic stroke minor 1 week, confirmed by cerebral imaging

Exclusion Criteria:

* severe aphasia (NIHSS criteria 9: sup or egal: 2)
* Chronic psychiatric preexistant desease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
acceptability | at 6 months
  Participation rate in the study

SECONDARY OUTCOMES:
Rates of anxiety and depression | at 3 and 6 months
  Montgomery and Asberg Depression Rating Scale(depressive patients) and wide COVI (anxious patients)
Evaluation of quality of life | at 3 and 6 months
  MM20-QOL scale
Evaluation of functional recovery | at 3 and 6 months
  * Barthel index and Rankin score
  * NIHSS score
Assessment of apathy | at 3 and 6 months
  apathy index
Categorization of patients | 6 months
  according to their pattern of coping with specific scales and RWCQ (Revised Ways of Coping Questionnaire - stroke modified version) QSSP (Questionnaire de soutien social perçu)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène MAHAGNE, PH, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU Nice, Nice, France